CLINICAL TRIAL: NCT05331248
Title: Training Leaders to Prevent and Reduce Domestic Violence in Their Communities: Experimental Evidence From Peru
Brief Title: Training Local Leaders to Prevent and Reduce Domestic Violence Evidence From Peru
Acronym: LIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Abdul Latif Jameel Poverty Action Lab (Other); Innovations for Poverty Action (Other); Medical Research Council, South Africa (Other); Inter-American Development Bank (Other); Wellspring Philanthropic Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0228; 1R01HD101581-01A1 (NIH); 14498 (Other: Innovations for Poverty Action)
Record Dates: First submitted 2022-02-16; First posted 2022-04-15 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Domestic Violence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- LIA Household Training (Experimental): This treatment arm is an 8-session training with a tailored schedule at the household level that targets couples at risk of domestic violence. The sessions are delivered by Community Health Volunteers: 1 Facilitator and 1 Community Agent. The training aims to raise awareness of IPV and social norms around domestic violence and is delivered at the household level in a private environment. Additionally, the intervention includes sessions on soft skills and conflict resolution. The session topics are: i) gender roles, beliefs and stereotypes; ii) violence, cultural patterns and human rights; iii) healthy relationships within the family; iv) good treatment between family members and self-care; v) Assertive communication; vi) resolution and conflict management; vii) resources for domestic violence cases; and viii) leadership and women's agency.
  Interventions: Behavioral: Leaders in Action: Household Treatment
- LIA Group Training (Experimental): This treatment arm is an 4-session training delivered in gender-segregated groups at the village level that targets couples at risk of domestic violence in separate spaces. The sessions are delivered by Community Health Volunteers: 1 Facilitator and 1 Community Agent. The training aims to raise awareness of IPV and social norms around domestic violence and is delivered at the household in a private environment. The sessions topics are: i) gender roles, beliefs and stereotypes; ii) violence, cultural patterns and human rights; iii) healthy relationships within the family; iv) good treatment between family members and self-care; v) assertive communication; vi) resolution and conflict management; vii) resources for domestic violence cases; and viii) leadership and women's agency.
  Interventions: Behavioral: Leaders in Action: Group Treatment
- LIA Household and Group Training (Experimental): This treatment arm combines LIA Household and Group training. Villages in this arm will first receive the 8-sessions household-level intervention, then the 4-sessions of village-level gender-segregated group intervention will follow. The session topics for both interventions are: i) gender roles, beliefs and stereotypes; ii) violence, cultural patterns and human rights; iii) healthy relationships within the family; iv) good treatment between family members and self-care; v) assertive communication; vi) resolution and conflict management; vii) resources for domestic violence cases; and viii) leadership and women's agency.
  Interventions: Behavioral: Leaders in Action: Household Treatment; Behavioral: Leaders in Action: Group Treatment
- Control group (No Intervention): Villages in the control group will not receive any intervention.

INTERVENTIONS:
Behavioral: Leaders in Action: Household Treatment — The Household Treatment (HT) followed a door-to-door delivery approach: CHVs, in coordination with the local Women Emergency Center (CEM), offered 8 treatment sessions to households in the targeted sample. The sessions took place over a period of 1 to 2 months at the residences of the female participants. This intervention was subject to a second-stage randomization to include edutainment videos in its implementation for the HT only treatment arm. In 31 randomly selected HT villages, all targeted households watched the edutainment component as part of the HT program, and in the other 31 HT villages, only 50% of the targeted households were randomly assigned to watch the edutainment component.
  Other Names: HT
  Arms: LIA Household Training; LIA Household and Group Training
Behavioral: Leaders in Action: Group Treatment — The group-based approach (Group Treatment, or GT) entailed 4 workshops involving various activities and group discussions. The group sessions directed at men had a slightly different curriculum than those directed at women, and always had at least one male CHV in the room facilitating the session. GT sessions took place over one month in each community in village community centers, schools, churches, or other communal spaces where village residents would often gather, and lasted for approximately two hours. The edutainment component was screened in every GT workshop.
  Other Names: GT
  Arms: LIA Group Training; LIA Household and Group Training

SUMMARY:
Leaders in Action (LIA) is a norms-centered intervention that aims to reduce the acceptance and prevent the incidence of Intimate Partner Violence (IPV) in Peru by shifting social norms. This project takes advantage of the randomization of LIA across 250 villages.

LIA has two delivery models: a household-based module (HT), consisting of household training sessions by Community Health Volunteers, and a group-based module (GT) with education sessions in small gender-segregated groups organized by trained facilitators. The investigators will cross-randomize each approach to assess efficiency in reducing domestic violence and changing social norms about tolerance toward violence and gender roles. The study disentangles the impact of the two modules separately, as well as the interaction of the modules, while explicitly addressing methodological concerns of previous studies: reporting bias from self-reported domestic violence, limited statistical power and lack of long-term effects measures.

Potential and actual victims of IPV may profit from the intimate atmosphere of household visits, and that on the side of women, the transmission of information about IPV and services for victims may be facilitated in more private settings. At the same time, group-level workshops about harmful gender stereotypes and gender norms for women should, through social interactions and norm change, reinforce the effects of household-level treatments for women. The experiment will shed light on the potential mechanisms at play and the theoretical framework underlying IPV through extensive data collection and the calculation of heterogeneous effects. The goal of this project is to deliver new rigorous evidence to the scientific and policy community by experimentally evaluating the impact of a state-run IPV intervention and its main components. It provides insights into the effectiveness of distinct program components, assesses cost-effectiveness as well as potential to scale, and evaluates the mechanisms leading to the reduction of IPV.

DETAILED DESCRIPTION:
Leaders in Action (LIA) is a norms-centered intervention run by the Peruvian Ministry for Women and Vulnerable Populations (MIMP) that aims to reduce the acceptance and incidence of Intimate Partner Violence (IPV) in Peru by shifting social norms. LIA has two main implementation phases: first, the recruitment of Community Health Volunteers (CHVs) and second, the delivery of content against IPV. The delivery of the intervention is assisted by MIMP professionals working in local "Women Emergency Centers" (Centro de Emergencia Mujer, or CEM), a nationwide network of hubs run by the MIMP that offer wide-ranging support services to IPV victims. The CEMs also implement other IPV prevention interventions at the local level.

CEM's Promotors (MIMP's professionals working at local CEM) recruit leaders of local social organizations and train them to be Facilitators of LIA. Facilitators are the principal CHVs located in each district center who conduct LIA activities. Another type of CHVs are leaders at the village-level who are trained by Facilitators to become Community Agents (CAs). Both CAs and Facilitators work together to conduct the second phase of LIA: the delivery of the intervention through its two delivery models, the Household Treatment (HT) and the Group Treatment (GT).

Originally, the study was designed to only evaluate the HT. Thus, a first randomization was conducted on our study sample with an even split of 125 control villages and 125 treatment villages. The research team and Innovations for Poverty Action (IPA) Peru deployed a census to identify the population of women in sample villages who met the eligibility criteria for the study, and conducted an in-depth baseline survey on women who reported IPV in the census. The implementation of the HT began in 2020, and was interrupted by the Covid-19 pandemic. The MIMP paused the program in March 2020 until national lockdowns were rescinded in February 2022. Given the intense migration and other demographic changes that took place during the 23-month interruption, as well as the potential for new IPV exposure over that period, new census and baseline surveys were conducted in 2022, which were used to define the final targeted sample for the intervention.

Our study tests two different delivery modes of the program, the HT and the GT, as well as their combination, in a cross-randomized design. The 250 villages in our study sample were randomized into 4 treatment arms following a factorial randomization model. This resulted in 62 villages receiving only the HT (HT only), 62 villages receiving only the GT (GT only), 63 villages receiving both the HT and GT (HT+GT), and 63 villages in the control group. The randomization procedure was stratified by CEM, the level of IPV risk, and the 2018 treatment status (villages that had begun implementation of the HT were restricted to remain in the HT only or HT+GT treatment arms).

The MIMP's original HT design followed a door-to-door delivery approach: CHVs, in coordination with the local CEM, offered 8 treatment sessions to households at risk of IPV. These HT sessions took place over a period of 1 to 2 months and were conducted in participants' residences. While all adult household members were invited to participate, the recipients of the HT were, in practice, primarily women. As a result, this delivery mode may have been ineffective at influencing norms and beliefs of male participants. The household-centered approach is also expensive and difficult to scale up. Thus, together with the MIMP, the research team developed modifications to the HT which resulted in the innovations described below.

First, in collaboration with the MIMP, the research team and IPA Peru developed a telenovela-style series as a key component of the LIA program (edutainment component). The series consists of four videos that reinforce themes of relationship conflict, masculinity, and social norms around gender. The edutainment component was randomized for the HT only treatment arm, so that in 31 villages, all households targeted for HT watched the edutainment component as part of the program, and in other 31 villages, only 50% of the households targeted for HT watched the edutainment component. In this second group, the households selected to watch the edutainment videos were randomly selected, which will allow the research team to experimentally identify the effect of the edutainment videos. In the other treatment arms (GT only and HT+GT), the edutainment component is implemented for all participants.

Second, in order to strengthen the effect of LIA and to reach potential perpetrators, which are predominantly men, as well as victims of IPV, we developed a different delivery format with the MIMP: the GT. The GT follows a gender-segregated yet community-wide delivery approach in a group discussion format. Existing evidence suggests that interventions which target both perpetrators and victims can have a substantial impact on attitudes towards and the incidence of IPV, and that simultaneously addressing IPV from different angles can be particularly effective (Chakraborty, P., Osrin, D. and Daruwalla, N., 2020; Abramsky, T. et al., 2014). These approaches commonly stress the importance of collaborative learning in support-group-style sessions to confront ideas of masculinity and gender norms. Moreover, norms change is more likely to happen when individuals are aware of relevant peers who are also changing their beliefs (Bursztyn, L., González, A. L., Yanagizawa-Drott, D. (2018)). As a result, the investigators proposed separating groups by gender to provide tailored settings during intervention.

* This group-based approach entailed 4 GT workshops that integrated various activities and group discussions focused on the same content as the HT. The group workshops directed at men had a slightly different curriculum than those directed at women, and always had at least one male CHV in the room facilitating the workshop. In order to meet this criteria during implementation, the MIMP required a larger number of male CHVs than those who were initially recruited through social organizations; men are usually recruited in disproportionately low numbers for this style of volunteer work, and the initial number of male CHVs was not sufficient for implementation of the GT. As a result, male CHVs were recruited as program Facilitators from local universities, communal associations, and other frequently-transited areas. GT sessions took place over the course of one month in village community centers, schools, churches, or other communal spaces where village residents would often gather, and lasted for approximately two hours. Larger villages held multiple GT sessions per workshop to cover all potential participants, and some villages were re-visited some months after the expected implementation time to ensure a high uptake.
* Participant targeting during the GT was the same as in other treatment arms: MIMP CHVs approached the houses of women in the targeted sample, and extended an invitation for them and their male partners to participate in the intervention. However, given that the GT is designed to involve the village community at large, invitations for the GT were extended to all adults in the village. Households in the targeted sample were approached door-to-door multiple times in the week before the GT session, while the rest of the village households were only approached once per workshop. Aside from door-to-door recruiting, the whole village received a notice an hour before each GT session through a loudspeaker usually used for other village-wide activities.
* The topics covered during both the HT and GT were equivalent to ensure comparability. These topics were: i) gender roles, beliefs and stereotypes; ii) violence, cultural patterns and human rights; iii) healthy relationships within the family; iv) respect between family members and self-care; v) assertive communication; vi) resolution and conflict management; vii) resources for domestic violence cases; and viii) leadership and women's agency.

Third, 50% of the villages assigned for either the HT only, GT only, or HT+GT treatment arms (94 villages total) were randomly selected to target one village leader (e.g. village president) to receive treatment given the village's treatment assignment. This will evaluate if community leaders are impactful in shifting norms at the village level.

Fourth, we randomized 50 percent of the treated villages to target a random selection of 30% of women who were interviewed in the census but did not report ever experiencing any form of IPV by their current partner. This will allow the research team to measure community-level impacts of the intervention through treatment density.

After the conclusion of both the HT and the GT, a set of qualitative interviews were conducted with the goal of informing the research team on the channels through which the treatments could be reducing IPV, as well as capturing information relevant to the design of the endline survey.

The research team plans to conduct an endline survey 6-months after the MIMP's implementation of the HT and GT to evaluate the impact of the LIA program and its different innovations on outcome measures such as: IPV, physical health, mental health, tolerance towards IPV, female agency, and social norms.

ELIGIBILITY:
Eligibility to receive the initial census: Women between the ages of 18-59 in 2022, who lived with a male partner, and who were permanent residents in villages from our sample (defined as living in the village for at least 4 months of the year).

Eligibility to be part of the targeted sample:

* Women identified to be at risk of suffering from IPV in the census, who as a result, also received a baseline survey.
* In 50 percent of the treatment villages chosen at random, an additional 30% of women randomly selected from the census.
* Male partners of women in the targeted sample.
* Across a sub-sample of 94 treatment villages chosen at random, 1 village leader. Specifically, we identified two village leaders, one male and one female, and randomly selected which of the genders was selected for targeting. This resulted in 50 women leaders and 44 men leaders, and their partners.

Eligibility for the endline survey sample:

* We plan to interview all men, women, and village leaders in our targeted sample.
* We will also interview 4 additional women per village who were eligible to receive the initial census but were not part of the targeted sample, as well as their male partners, to measure spillover effects.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8754 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Women's Reporting of Intimate Partner Violence | 06 months after the intervention
  For women only. The researchers will replicate a standard Demographic Household Survey domestic violence module, administered through a self-paced ballot-style questionnaire. The indicator will take the value of 1 if a woman reports at least 1 event of intimate-partner violence, and 0 if a woman reports not having experienced any events of intimate-partner violence. The indicator values are 0 and 1; with 1 meaning a woman suffered from intimate-partner violence and 0 meaning a woman did not suffer intimate-partner violence in the reporting period.
Women's Index of Physical Health | 06 months after the intervention
  For women only. The researchers will use World Health Organization questionnaires on physical health. The index values are 0 to 1; higher scores mean better outcomes.
Women's Index of Mental Health | 06 months after the intervention
  For women. The researchers will use questions from the Kessler Psychological Distress Scale 6 (K6) for mental distress. The index values are 0 to 1; higher scores mean better outcomes.
Men's Index of Mental Health | 06 months after the intervention
  For men. The researchers will use questions from the Kessler Psychological Distress Scale 6 (K6) for mental distress. The index values are 0 to 1; higher scores mean better outcomes.
Men's Index of Tolerance towards Violence against Women | 06 months after the intervention
  For men. The researchers will use 9 statements about the justification of violence (asking whether the participants agree or disagree with these statements). The index values are 0 to 1; higher scores mean worse outcomes.
Women's Index of Tolerance towards Violence against Women | 06 months after the intervention
  For women. The researchers will use 9 statements about the justification of violence (asking whether the participants agree or disagree with these statements). The index values are 0 to 1; higher scores mean worse outcomes.

SECONDARY OUTCOMES:
Women's Index of Agency | 06 months after the intervention
  For women only. The researchers will use 3 items of a self-efficacy scale. The scale values are 0 to 1; higher scores mean better outcomes.
Men's Index of Social Norms | 06 months after the intervention
  For men. The researchers will use 6 statements about gender roles and norms statements about the justification of violence (asking whether the participants agree or disagree with these statements). The index values are 0 to 1; higher scores mean better outcomes.
Women's Index of Social Norms | 06 months after the intervention
  For women. The researchers will use 6 statements about gender roles and norms (asking whether the participants agree or disagree with these statements). The index values are 0 to 1; higher scores mean better outcomes.
Women's reporting of Violence from non-Partner | 06 months after the intervention
  For women only. The researchers will replicate standard Demographic Household Survey questions for non-partner violence, administered through a self-paced questionnaire. The indicator will take the value of 1 if a woman reports at least 1 event of non-partner violence, and 0 if a woman reports not having experienced any events of non-partner violence. The indicator values are 0 and 1; with 1 meaning a woman suffered from non-partner violence and 0 meaning a woman did not suffer non-partner violence in the period.
Men's reporting of Intimate Partner Violence | 06 months after the intervention
  For men only. The researchers will replicate some sections from the Demographic Household Survey domestic violence module, administered through a self-paced ballot-style questionnaire. Researchers will limit the questions asked about violence experienced to psychological IPV only when surveying men. The indicator will take the value of 1 if the man reports at least 1 event of psychological intimate-partner violence, and 0 if a man reports not having experienced any events of psychological intimate-partner violence. The indicator values are 0 and 1; with 1 meaning a man suffered from psychological intimate-partner violence and 0 meaning a man did not suffer psychological intimate- partner violence in the reporting period.

CONTACTS AND LOCATIONS:
Overall Officials: Erica Field, PhD, Principal Investigator — Duke University; Livia Schubiger, PhD, Principal Investigator — University of Oxford; Ursula Aldana, PhD, Principal Investigator — Instituto de Estudios Peruanos
Locations (1):
- Innovations for Poverty Action, Lima, Peru

REFERENCES:
- [Background] Ellsberg M, Arango DJ, Morton M, Gennari F, Kiplesund S, Contreras M, Watts C. Prevention of violence against women and girls: what does the evidence say? Lancet. 2015 Apr 18;385(9977):1555-66. doi: 10.1016/S0140-6736(14)61703-7. Epub 2014 Nov 21. PMID 25467575
- [Background] Chakraborty P, Osrin D, Daruwalla N. "We Learn How to Become Good Men": Working with Male Allies to Prevent Violence against Women and Girls in Urban Informal Settlements in Mumbai, India. Men Masc. 2020 Aug;23(3-4):749-771. doi: 10.1177/1097184X18806544. Epub 2018 Oct 18. PMID 32903823
- [Background] Abramsky T, Devries K, Kiss L, Nakuti J, Kyegombe N, Starmann E, Cundill B, Francisco L, Kaye D, Musuya T, Michau L, Watts C. Findings from the SASA! Study: a cluster randomized controlled trial to assess the impact of a community mobilization intervention to prevent violence against women and reduce HIV risk in Kampala, Uganda. BMC Med. 2014 Jul 31;12:122. doi: 10.1186/s12916-014-0122-5. PMID 25248996